CLINICAL TRIAL: NCT00455455
Title: Corneal and Conjunctival Sensitivity and Staining Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Craig Woods, Research Manager, Centre for Contact Lens Research
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P/245/06/L
Record Dates: First submitted 2007-03-23; First posted 2007-04-03 (Estimated); Results first posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-06

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optifree RepleniSH Multipurpose Disinfecting Solution (Active Comparator)
  Interventions: Drug: Optifree RepleniSH Multipurpose Disinfecting Solution
- ReNu Multiplus Multipurpose Solution (Active Comparator)
  Interventions: Drug: ReNu Multiplus Multipurpose Solution

INTERVENTIONS:
Drug: Optifree RepleniSH Multipurpose Disinfecting Solution — lens care system
  Other Names: lens care system
  Arms: Optifree RepleniSH Multipurpose Disinfecting Solution
Drug: ReNu Multiplus Multipurpose Solution — lens care system
  Other Names: lens care system
  Arms: ReNu Multiplus Multipurpose Solution

SUMMARY:
The primary objective of this study is to compare subjective symptoms and ocular health in a group of individuals who are currently wearing soft contact lenses on a daily wear basis, after a short period of no lens wear and during the time course when using differing care regimens.

DETAILED DESCRIPTION:
The primary objective of this study is to compare subjective symptoms and ocular health in a group of individuals who are currently wearing soft contact lenses on a daily wear basis, after a short period of no lens wear and during the time course when using differing care regimens. Observations will be made to monitor physiology.

ELIGIBILITY:
Inclusion Criteria:

An eligible participant is one who:

* Is between 17-45 years old and has full legal capacity to volunteer.
* Has read and signed an information consent letter, after having the opportunity to ask questions and receive acceptable answers.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Does not experience any dryness related symptoms during lens wear (i.e. at least 12 hours of comfortable wearing time)
* Is correctable to a visual acuity of 6/7.5 (20/25) or better (each eye) with their habitual vision correction.
* Has normal binocular vision (no strabismus, no amblyopia).
* Has clear corneas and no active ocular disease.
* Has had an ocular examination in the last two years. Has a distance contact lens prescription between +0.50D to +6.00 DS and -0.50D and -12.00 DS.
* Has astigmatism less than or equal to -1.00DC.
* Agrees to wear the study lenses on a daily wear basis.
* Has a pair of glasses with updated prescription and agrees to wear them during the period no lens wear (7-10 days) as required by the study.

Exclusion Criteria:

A person is ineligible if he/she:

* Has undergone corneal refractive surgery.
* Is aphakic.
* Has any active ocular disease.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that may affect ocular health.
* Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study.
* Is pregnant or lactating.
* Is participating in any other clinical or research study.
* Has a known clinically significant sensitivity to the contact lens care solutions used in the study.
* Has ocular or systemic allergies that could adversely affect contact lens wear.
* Currently wears lenses on a continuous or extended wear basis.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
* Has pinguecula/pterygium that, in the investigator's judgment, makes contact lens wear inadvisable.
* Is a rigid lens wearer.
* Has corneal staining graded as 2 (macropunctate) or greater in any corneal region in either eye, sum of corneal staining type (severity) of greater than or equal to 4 across the entire cornea in either eye, or any corneal staining covering greater than or equal to 20% in any corneal region in either eye.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, M.Optom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, School of Optometry, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Situ P, Simpson TL, Jones LW, Fonn D. Effects of silicone hydrogel contact lens wear on ocular surface sensitivity to tactile, pneumatic mechanical, and chemical stimulation. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6111-7. doi: 10.1167/iovs.09-4807. Epub 2010 Jun 30. PMID 20592230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from local communities in Kitchener-Waterloo, Canada between May 2007 and Feb 2008.
Pre-assignment Details: 64 participants recruited and screened; 14 withdrawn prior to the group assignment due to loss of interest, relocation and inconvenience.
Groups:
- RepleniSH First, Then ReNu: Following a washout period, use RepleniSH for lens care in first period and ReNu in second period (after the second washout period)
- ReNu First, Then RepleniSH: Following a washout period, use ReNu for lens care in first period and RepleniSH in second period (after the second washout period)
Period: Washout
Arm/Group | RepleniSH First, Then ReNu | ReNu First, Then RepleniSH
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: First Intervention
Arm/Group | RepleniSH First, Then ReNu | ReNu First, Then RepleniSH
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0
Period: Washout
Arm/Group | RepleniSH First, Then ReNu | ReNu First, Then RepleniSH
Started | 25 | 24
Completed | 24 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | RepleniSH First, Then ReNu | ReNu First, Then RepleniSH
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Group: includes groups randomized to use RepleniSH in the 1st period and ReNu in the 2nd period, and first use ReNu and use RepleniSH in the second period.
Arm/Group | Entire Study Group
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15
Region of Enrollment [Number; unit: participants]
  Canada | 50

OUTCOME MEASURES:

1. Primary Outcome: Corneal Sensitivity
Description: The detection threshold, the lowest level at which a stimulus to the cornea in a unit of percent CO2 can be detected was measured. Sensitivity is the reciprocal of the detection threshold.
Time Frame: baseline
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: percent CO2
Groups:
- RepleniSH: use RepleniSH for lens care in either first period or second period
- ReNu: Use ReNu for lens care in either first period or second period
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
percent CO2 | 26.9 (13.0) | 25.5 (12.9)

2. Secondary Outcome: Corneal Staining Grade
Description: A 0-100 grading scale based on the extent of corneal staining (0 none, 100 full area).
Time Frame: baseline
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
units on a scale | 1.3 (2.0) | 1.8 (3.0)

3. Primary Outcome: Corneal Sensitivity
Description: as for outcome 1
Time Frame: day 7
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: percent CO2
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
percent CO2 | 25.5 (13.4) | 22.1 (13.8)

4. Secondary Outcome: Corneal Staining Grade
Description: A 0-100 grading scale based on the extent of corneal staining (0 none, 100 full area).
Time Frame: day 7
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
units on a scale | 4.7 (7.5) | 49.9 (39.9)

5. Primary Outcome: Conjunctival Sensitivity
Description: The detection threshold, the lowest level at which a stimulus to the conjunctiva in a unit of percent CO2 can be detected was measured. Sensitivity is the reciprocal of the detection threshold.
Time Frame: baseline
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: percent CO2
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
percent CO2 | 48.7 (20.2) | 49.6 (18.7)

6. Primary Outcome: Conjunctival Sensitivity
Description: as for outcome 5
Time Frame: day 7
Population: intent to treat analysis including only participants who had completed the study
Measure: Mean (Standard Deviation); unit: percent CO2
Groups:
- RepleniSH: use RepleniSH for lens care in the first period and the second period
- ReNu: use ReNu for lens care in the first period or the second period
Arm/Group | RepleniSH | ReNu
Number analyzed (Participants) | 48 | 48
percent CO2 | 50.5 (20.2) | 46.2 (22.4)

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no adverse events
Arm/Group | RepleniSH | ReNu
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

LIMITATIONS AND CAVEATS:
Sample size completed as anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No